CLINICAL TRIAL: NCT06508177
Title: Does Postoperative Analgesic Modalities Effect Blood Creatin Phosphokinase Levels After Laparoscopic Cholecystectomy Surgery?
Brief Title: CPK Levels After LC and Association With Analgesic Modalities
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SamsunU_LapCholecyst_CK
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Myotoxicity
Keywords: creatine phosphokinase; cholecystectomy; interfascial plane blocks
MeSH Terms: conditions — Myotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interfascial plane blocks: Patients who are preferred to apply interfascial plane blocks as part of multimodal analgesia in the postoperative analgesia plan will be evaluated in this group.
  Interventions: Other: İnterfascial plane block; Other: Standart analgesia plan
- Control: Multimodal analgesia plans that does not include interfascial plane blocks
  Interventions: Other: Standart analgesia plan

INTERVENTIONS:
Other: İnterfascial plane block — Interfascial plane blocks will be added to the routine analgesia plan as part of multimodal analgesia.
  Groups: Interfascial plane blocks
Other: Standart analgesia plan — This is the routine analgesia plan applied in our clinic.

SUMMARY:
Regional anesthesia and analgesia technics are widely and securely used during general surgery procedures. Interfascial plane blocks are the latest used ones for analgesia. There are studies in literature indicating that bupivacaine cause myotoxicity. The investigators aimed to examine plasma creatine phosphokinase (CPK) levels to see whether myotoxicity occurs or not after fascial plane blocks are applied to patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
During 3 months period all elligible patients undergoing laparoscopic cholecystectomy surgery will be included in the study. Different postoperative analgesic modalities will be used according to the anesthesists experience. During routine blood sample tests plasma creatin phosphokinase (CPK) levels will be tested 3 times of all patients(preoperative, postoperative 6th hour, postoperative 24th hour). Data will be analysed and patients will be grouped according to the analgesic modalities used.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Laparoscopic cholecystectomy
* under General Anesthesia

Exclusion Criteria:

* Morbidly obesity or cachexia
* local anesthetic allergies
* myopathies
* coagulopathies
* Obstructive sleep apne syndrome
* hearth diseases
* liver diseases
* kidney diseases
* thyroid-parathyriod dieseas
* hiperlipidemias using Statins(HMG-CoA reductase inhibitors)
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent laparoscopic cholecystectomy ASA 1-3. age:18-70
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
CPK levels | at postoperative 24th hour
  Serum creatine phosphokinase levels at 24th hour

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Study Chair — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rakhi V, Kaushal S, Singh S. Measurement of bupivacaine induced myotoxicity in interfascial plane blocks: A randomised controlled trial. Indian J Anaesth. 2021 Dec;65(12):886-891. doi: 10.4103/ija.ija_848_21. Epub 2021 Dec 22. PMID 35221361